CLINICAL TRIAL: NCT03233087
Title: Diagnosis and Prognosis for Aortic Aneurysm aNd Dissection in Anzhen
Brief Title: Diagnosis and Prognosis for Aortic Aneurysm aNd Dissection in Anzhen(DPANDA) Study
Status: Recruiting | Type: Observational
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Beijing Luhe Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); The First Hospital of Jilin University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The General Hospital of Northern Theater Command (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: DPANDA
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Aortic Aneurysm; Aortic Dissection
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Top third of subjects based levels of selected biomarker.
- Middle third of subjects based levels of selected biomarker.
- Bottom third ofsubjects based levels of selected biomarker.

SUMMARY:
The registry study aims to determine serial biomarkers to diagnosis and prognosis of aortic aneurysm/aortic dissection.

DETAILED DESCRIPTION:
The study aims to investigate the role of candidate biomarkers in the diagnosis and prognosis of AA and AD. In the diagnosis part, we begin with a discovery phase where individually matched case-control study. Patients within each disease outcomes (i.e. AD, AMI, PE, AA without AD and healthy controls) are age and sex matched and retrospectively included.In the prognosis part of the study, patients with confirmed AA and AD are enrolled. The primary outcome is the all-cause mortality based on the death certificates. The secondary outcome is the in-hospital mortality according to the patients'medical records.

ELIGIBILITY:
Inclusion Criteria:

Retrospective

* All patients who were referred to the surgical service for evaluation and management of aortic dissection were included.

Perspective

* Patients with initial suspicion of having AAD were perspectively enrolled.

Exclusion Criteria:

Retrospective

* Patients who received packed red blood cells, whole blood, or platelets less than 10 days before the blood sample was taken;
* Patients with aortic trauma, pseudo aneurysm, history of heart failure, renal dysfunction, severe pulmonary diseases, or active cancer;
* Patients who entered the hospital for checkups after surgery.

Perspective

* Patients in whom there is little or no suspicion of a life-threatening disease;
* Patients with confirmed acute myocardial infarction,angina or pulmonary embolism
* The symptoms were clearly not related to AD (e.g. pleurisy, pneumonia, acute abdominal diseases).

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: These cohorts consist of patients who was diagnosed as thoracic aortic aneurysm/dissection or initial suspicion of having thoracic aortic aneurysm/dissection.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dignosis of each participant | These data is collected from the cases' medical record in an average of 6 month after the sample recruiting
  1. Patients with Aneurysm/Dissection had image information from ultrasound cardiograms and computed tomography to confirm the final diagnosis.
  2. AMI if they had chest pain lasting >20 min, diagnostic serial ECG changes comprising new pathological Q waves or ST-segment and T-wave changes, and a plasma creatine kinase-MB elevation greater than twice the normal level or cardiac troponin I (cTnI) level greater than 0.1 ng/mL.
  3. Diagnosis of PE was confirmed by positive spiral computed tomography or pulmonary angiography, a high probability on ventilation perfusion scintigraphy, or a proximal deep vein thrombosis documented on compression ultrasonography or angiography.
Prognosis of each participant | These data is collected from the cases' medical record or during follow-up visit at 2-4 years after discharge.
  Prognosis information including all-cause mortality and in-hospital mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China